CLINICAL TRIAL: NCT05422859
Title: Mobile and Digital Application in Heart Failure Networks Berlin/Brandenburg
Acronym: MobiDig
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Heart Institute (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Principal Investigator, Sabine Huebler, Head of Studienzentrale, German Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MobiDig
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MobiDig (Other): 50 patients will have access to a mobile phone application for 3 months.
  Interventions: Other: MobiDig

INTERVENTIONS:
Other: MobiDig — The application will contain the following modules:
  1. information and knowledge about heart failure;
  2. vital sign diary, which can be sent to the certified HFU
  3. pedometer (individualized step-goal), cardiac home training videos
  4. "frequently asked questions" and connection to a certified HFU provider by a heart failure hotline

SUMMARY:
The MobiDig trial is designed to evaluate an implementation of a mobile phone application with secondary preventive/rehabilitative modules for patients with heart failure in certified Heart Failure Unit centers in Berlin and Brandenburg.

The aim is to evaluate the effect on quality of life, symptoms and the course of the disease. In addition, the acceptance, adherence and user behavior as well as the implementation potential for a permanent introduction of the application in national heart failure networks will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of heart failure
* Treatment in a certified Heart Failure Unit center in Berlin or Brandenburg
* Written informed consent of the participants
* User of a mobile device with an iOS operating system

Exclusion Criteria:

* Addiction or other illnesses that do not allow the participants to assess the nature and scope as well as possible consequences of participation or its scientific evaluation
* insufficient knowledge of the German language, which is necessary to use the application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance of the application | 3 months
  The acceptence of the application will be measured by the User Experience Questionnaire. It consists of 9 items that can be rated on a 7-point Likert scale. -3 (fully agree with negative term) to +3 (fully agree with positive term). A higher total score means a better outcome.
Change in quality of life | Baseline and 3 months
  Quality of life measured by Kansas City Cardiomyopathy Questionnaire using the validated 12-item version which has been described by Spertus et Jones (doi: 10.1161/CIRCOUTCOMES.115.001958.) A higher score means a better outcome.
Patient reported outcomes | Baseline and 3 months
  Health-related quality of life will be measured by the "Patient Related Outcome and Measurement Information System" (PROMIS) test. Including 23 items that will be analyzed via Likert scale 1 (impossible/never) to 5 (no limitations/very good). A higher score means a better outcome.
Change in symptoms of heart failure | Baseline and 3 months
  Symptoms of heart failure will be assessed by the New York Heart Association functional class. Consisting of four classes (I-IV), the higher, the worse the outcome.
Change in six-minute walk distance | Baseline and 3 months
  Functional capacity will be assessed by the 6-minute walk test
Change in daily walking distances | Baseline and 3 months
  Functional capacity will be assessed by the steps taken within 24 hours (pedometry).
Change in heart failure biomarker | Baseline and 3 months
  Heart failure severity will be assessed by the biomarker NT-proBNP.
Number of hospitalizations | 3 months
  Number of hospitalizations for heart failure will be assessed.
Length of hospitalizations | 3 months
  Length of in-hospital stay of hospitalizations for heart failure will be assessed.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Deutsches Herzzentrum der Charité - Universitätsmedizin Berlin, Berlin, Deutschland
  - Charité - Universitätsmedizin Berlin: Campus Virchow-Klinikum, Berlin
  - Herzzentrum Berlin, Bernau

IPD SHARING:
Plan to Share IPD: No